CLINICAL TRIAL: NCT00998634
Title: Randomized, Placebo-controlled Trial to Test Safety, Tolerability and Efficacy of Lithium Carbonate in Spinocerebellar Ataxia 2
Brief Title: Safety and Tolerability of Lithium in Spinocerebellar Ataxia 2 (SCA2)
Acronym: LISCA2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Alessandro Filla, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCA_LITIO_12; EUDRACT N°2009-016317-20
Record Dates: First submitted 2009-10-16; First posted 2009-10-20 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: SPINOCEREBELLAR ATAXIA 2
Keywords: SCA2; Lithium
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LITHIUM CARBONATE 150 and/or 300 mg (Experimental)
  Interventions: Drug: LITHIUM CARBONATE
- PLACEBO (Placebo Comparator)
  Interventions: Drug: LITHIUM CARBONATE

INTERVENTIONS:
Drug: LITHIUM CARBONATE — Lithium Carbonate will be dosed based on lithiemy, which will be in the range 0.9-1.2 mEq/L. Maximum allowed dose will be 1500mg/day.

SUMMARY:
The purpose of this study is to determine safety and tolerability of the treatment with lithium in Spinocerebellar Ataxia 2. Moreover, clinical symptoms, neuronal loss, quality of life and depressive symptoms, will be considered to further investigate the effect of lithium therapy.

DETAILED DESCRIPTION:
Patients will be progressively enrolled in the study and undergo a screening visit to test for inclusion/exclusion criteria. Patients will then be randomized to receive either Lithium carbonate or placebo. Patients will visit study center at 2, 4, 8, 12, 24, 36 and 48 weeks, for endpoint and laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of SCA2 (≥34 CAG in the ataxin-2 gene)
* Age ≥18, <80
* SARA score ≥8

Exclusion Criteria:

* SARA score >32
* Heart failure
* Liver disease
* Kidney failure
* Thyroid disease
* Sick sinus syndrome and/or significant ECG alterations
* Hyposodemia
* Treatment with diuretics
* Treatment with haloperidol and/or other antipsychotics
* Treatment with NSAIDs or corticosteroids
* Treatment with ACE inhibitors
* Treatment with aminophyllines
* Treatment with mannitol
* Pregnancy and/or breastfeeding
* Acute diseases that might interfere with the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Primary endpoint of the study will be the difference in the number and frequency of Severe Adverse Events (SAE) and Non Severe Adverse Events (nSAE) recorded during the study, between treatment and placebo group. | the endpoint will be recorded at all visits
  Adverse events and Severe Adverse events will be recorded during the trial at each visit starting from Baseline to Visit 8 at 48 weeks of treatment.

SECONDARY OUTCOMES:
Secondary outcome will be the Scale for the Assessment and Rating of Ataxia (SARA). Statistical analysis will be performed to compare the effect of treatment on both groups. | 0 weeks
Micro- and macrostructural Magnetic Resonance parameters will be compared before and after treatment. This will include Voxel Based Morphometry, resting functional MRI, Diffusion tensor imaging and MRI spectroscopy. | 0 weeks
The effect of Lithium on mood will be explored with the Beck depression inventory. | 0 weeks
Effect of Lithium on quality of life will be assessed with the EQ-5D scale. | 0 weeks
Secondary outcome will be the Scale for the Assessment and Rating of Ataxia (SARA). Statistical analysis will be performed to compare the effect of treatment on both groups. | 24 weeks
Secondary outcome will be the Scale for the Assessment and Rating of Ataxia (SARA). Statistical analysis will be performed to compare the effect of treatment on both groups. | 48 weeks
Micro- and macrostructural Magnetic Resonance parameters will be compared before and after treatment. This will include Voxel Based Morphometry, resting functional MRI, Diffusion tensor imaging and MRI spectroscopy. | 48 weeks
The effect of Lithium on mood will be explored with the Beck depression inventory. | 24 weeks
The effect of Lithium on mood will be explored with the Beck depression inventory. | 48 weeks
Effect of Lithium on quality of life will be assessed with the EQ-5D scale. | 24 weeks
Effect of Lithium on quality of life will be assessed with the EQ-5D scale. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Filla, MD, Principal Investigator — University Federico II
Locations (1):
- Dipartimento di Scienze Neurologiche, Napoli, Italy

REFERENCES:
- See also: University Federico II — http://www.unina.it
- See also: AOU Policlinico "Federico II" — http://www.policlinico.unina.it